CLINICAL TRIAL: NCT00436319
Title: Effect of the Duration of GnRH-analogue Downregulation on Pregnancy Rates in IVF
Brief Title: Duration of GnRH-analogue Downregulation and Pregnancy Rates
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHR-2
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: Infertility, downregulation, stimulation, agonists, long
MeSH Terms: conditions — Infertility

ARMS (2):
- 1 (No Intervention): In the control group (group 1) the initiation of the ovarian stimulation will be realized according to the typical long luteal protocol, two weeks after the initiation of the GnRH agonist administration.
- 2 (Other): In the study group (group 2) the initiation of the ovarian stimulation will be effectuated on the second day of the menstrual period.
  Interventions: Procedure: Duration of GnRH agonist downregulation

INTERVENTIONS:
Procedure: Duration of GnRH agonist downregulation — This is a randomized controlled trial. Patients will be randomized to two groups during the first consultation. GnRH agonist will be administrated according to the long luteal protocol. Down-regulation of the pituitary will be controlled on the first day of the menstrual period.
  The purpose of this study is to compare the pregnancy rates between the two groups. In the eventuality that pituitary down-regulation has not been confirmed (down-regulation levels determined as Ε2<80 pg/ml and progesterone <1.6 ng/ml), the patient will be assigned to a third group (group 3) and ovarian stimulation will only be initiated after down-regulation has been confirmed.
  The GnRH agonist that will be administrated is Buserelin Acetate. Recombinant FSH will be used for the ovarian stimulation and dose determination will be based on patient characteristics and previous history.
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether the probability of pregnancy is dependent on the duration of GnRH agonist downregulation in IVF cycles.

DETAILED DESCRIPTION:
GnRH agonists have been used extensively in assisted reproduction technologies for inhibition of gonadotropin secretion from the pituitary prior to initiation of ovarian stimulation. Administration of GnRH agonists results in the prevention of spontaneous LH surges, which lead to luteinization of the developing follicles, initiation of final oocyte maturation and a decrease in pregnancy rates.

GnRH agonists are usually administered according to two protocols: the short and long protocol.In the long protocol, downregulation with GnRH agonists is initiated either in the middle of the secretory phase, or at the beginning of the follicular phase. Stimulation of the ovaries with gonadotropins is initiated when downregulation is confirmed.

Administration of gonadotropins is usually started during the second or third week of treatment with GnRH agonists.The possibility of earlier initiation of the ovarian stimulation, if downregulation is confirmed at an earlier stage, has not been examined so far.

The purpose of this study is to assess whether the duration of pituitary downregulation with GnRH agonists, prior to initiation of ovarian stimulation with gonadotropins, has any effect on pregnancy rate, in women undergoing IVF.

ELIGIBILITY:
Inclusion Criteria:

* age under 39
* less than 3 previous IVF cycles
* BMI 18-29
* normal ultrasound of internal genital organs

Exclusion Criteria:

* polycystic ovarian syndrome
* endometriosis

Ages: 19 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-05; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Basil C Tarlatzis, MD PhD, Principal Investigator — Unit of Human Reproduction, 1st Department of Obst & Gyn, Aristotle University of Thessaloniki, Papageorgiou Hospital, Greece
Locations (1):
- Unit of Human Reproduction, 1st Department of Obst & Gyn, Aristotle University of Thessaloniki, Papageorgiou Hospital, Greece, Thessaloniki, Greece

REFERENCES:
- [Background] Damario MA, Moomjy M, Tortoriello D, Moy F, Davis OK, Rosenwaks Z. Delay of gonadotropin stimulation in patients receiving gonadotropin-releasing hormone agonist (GnRH-a) therapy permits increased clinic efficiency and may enhance in vitro fertilization (IVF) pregnancy rates. Fertil Steril. 1997 Dec;68(6):1004-10. doi: 10.1016/s0015-0282(97)00392-0. PMID 9418688
- [Background] Kolibianakis EM, Papanikolaou EG, Camus M, Tournaye H, Van Steirteghem AC, Devroey P. Menstruation-free interval and ongoing pregnancy in IVF using GnRH antagonists. Hum Reprod. 2006 Apr;21(4):1012-7. doi: 10.1093/humrep/dei415. Epub 2005 Dec 8. PMID 16339166